CLINICAL TRIAL: NCT01494649
Title: A Pilot Clinical Study Investigating the Efficacy of a Toothpaste in Providing Immediate and Short Term Relief From Dentinal Hypersensitivity
Brief Title: Pilot Study to Investigate the Efficacy of a Toothpaste in Providing Relief From Dentinal Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z7871335
Record Dates: First submitted 2011-09-01; First posted 2011-12-19 (Estimated); Results first posted 2013-05-08 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2012-08

CONDITIONS: Dentinal Sensitivity; Hypersensitivity
Keywords: dentinal; hypersensitivity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Toothpaste containing 0.454% stannous fluoride (Active Comparator): USA marketed toothpaste [test]
  Interventions: Drug: Test Toothpaste
- Toothpaste containing 0.76% sodium monofluorophosphate (Other): USA marketed toothpaste [negative control]
  Interventions: Drug: Negative Control Toothpaste

INTERVENTIONS:
Drug: Test Toothpaste — 0.454% stannous fluoride toothpaste
  Arms: Toothpaste containing 0.454% stannous fluoride
Drug: Negative Control Toothpaste — 0.76% sodium monofluorophosphate toothpaste
  Arms: Toothpaste containing 0.76% sodium monofluorophosphate

SUMMARY:
A pilot study to determine the ability of a stannous fluoride containing toothpaste to provide immediate and short term relief from dentine Hypersensitivity compared to a control toothpaste.

ELIGIBILITY:
Inclusion:

* Self-reported history of dentinal hypersensitivity lasting more than 6 months and less than 10 years
* Teeth showing signs of facial/cervical gingival recession and/or signs of erosion or abrasion.
* Teeth having a gingival index score of less than or equal to 1
* Teeth with a clinical mobility less than or equal to 1
* sensitive teeth from those meeting the EAR, GI and mobility criteria at screening, with sensitivity as measured by tactile stimulus (Yeaple probe, tactile threshold 10g) and evaporative (air) stimulus (Schiff Sensitivity Score ≥ 2).

Exclusion:

* Presence of chronic debilitating disease which could affect study outcomes.
* Any condition which causes xerostomia.
* Dental prophylaxis within 4 weeks of screening.
* Tongue or lip piercing or presence of dental implants.
* Professional desensitising treatment within 12 weeks of screening.
* Gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of screening, scaling or root planning within 3 months of screening.
* Teeth bleaching within 12 weeks of screening.
* Tooth with evidence of current or recent caries, or reported treatment of decay in 12 months of screening.
* Tooth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, teeth with full crowns or veneers, orthodontic bands or cracked enamel. Sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine, or not expected to respond to treatment with an over-the counter dentifrice.
* Daily doses of a medication which could interfere with the perception of pain.
* Currently taking antibiotics or have taken antibiotics within 2 weeks of baseline.
* Individuals who require antibiotic prophylaxis for dental procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2011-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- BioSci Research America, Inc., Las Vegas, Nevada, United States

REFERENCES:
- [Derived] Parkinson CR, Hughes N, Hall C, Whelton H, Gallob J, Mason S. Three randomized clinical trials to assess the short-term efficacy of anhydrous 0.454% w/w stannous fluoride dentifrices for the relief of dentin hypersensitivity. Am J Dent. 2016 Feb;29(1):25-32. PMID 27093773

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site
Groups:
- Test: Commercially available toothpaste containing 0.454% stannous fluoride, 1 inch strip brushed on each of the 2 selected sensitive teeth for 30 seconds, followed by thorough brushing of all teeth for at least 1 minute for 14 days twice daily.
- Negative Control: Toothpaste containing 0.76% sodium monofluorophosphate, 1 inch strip brushed on all teeth in the whole mouth for at least 1 minute for 14 days twice daily
Period: Overall Study
Arm/Group | Test | Negative Control
Started | 59 | 59
Completed | 59 | 58
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test | Negative Control | Total
Number analyzed (Participants) | 59 | 59 | 118
Age Continuous [Mean (Standard Deviation); unit: Years] | 35.7 (10.65) | 37.0 (9.98) | 36.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 74
  Male | 22 | 22 | 44
Region of Enrollment [Number; unit: Participants]
  USA | 59 | 59 | 118

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Tooth Hypersensivity to Air Stimuli Immediately Following Treatment
Description: Response to a constant (duration, pressure, temperature, distance from target) jet of air applied to a hypersensitive tooth was evaluated using Schiff Cold Air Sensitivity Scale. According to this analog scale hypersensitivity scores for the stimulated tooth is 0, 1, 2 or 3 (lower the score, lower the hypersensitivity).0= no response; 1= response and no discontinuation request; 2= response and discontinuation request; 3= painful response and discontinuation request. Change was calculated as Schiff score immediately after treatment minus Schiff score at baseline.
Time Frame: Baseline and immediately after treatment administration
Population: Intent to treat (ITT) population: All participants who were randomized, receive at least one dose of treatment, and had at least one post baseline efficacy evaluation. No data was imputed in the case of dropouts or missing data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Test: Commercially available toothpaste containing 0.454% stannous fluoride, 1 inch strip brushed on each of the 2 selected sensitive teeth for 30 seconds, followed by thorough brushing of all teeth for at least 1 minute for 14 days twice daily. The test product is a commercially available product.
Arm/Group | Test | Negative Control
Number analyzed (Participants) | 59 | 59
units on a scale | -0.42 [-0.53 to -0.30] | -0.32 [-0.43 to -0.21]
Statistical Analysis 1: Comparison: Test vs Negative Control; Null hypothesis is no difference between treatments. Tests were 2-sided; Test type: Superiority or Other; p = 0.2294, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; The model included treatment as a fixed factor and basline Schiff score as a covariate; Adjusted mean difference = -0.10, 95% CI 2-sided [-0.26 to 0.06] — Difference was calculated as adjusted mean change from baseline in 0.454% stannous fluoride toothpaste minus 0.76% sodium fluoride toothpaste. Negative difference favoured stannous fluoride toothpaste

2. Secondary Outcome: Adjusted Mean Change From Baseline in Tooth Hypersensitivity to Air Stimuli at Day 3
Description: Response to a constant (duration, pressure, temperature, distance from target) jet of air applied to a hypersensitive tooth evaluated using Schiff Cold Air Sensitivity Scale. According to this analog scale hypersensitivity scores for the stimulated tooth is 0, 1, 2 or 3 (lower the score, lower the hypersensitivity). 0=No participant response to stimulus, 1=responds but will continue, 2=responds and moves or requests discontinuation, 3=Painful response to stimulus, discontinuation requested. Change was Schiff score on Day 3 minus Schiff score at baseline.
Time Frame: Baseline and Day 3
Population: ITT population: All participants who were randomized, receive at least one dose of treatment, and had at least one post baseline efficacy evaluation. No data was imputed in the case of dropouts or missing data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Test | Negative Control
Number analyzed (Participants) | 59 | 58
units on a scale | -0.57 (0.515) [-0.69 to -0.44] | -0.45 (0.478) [-0.57 to -0.32]
Statistical Analysis 1: Comparison: Test vs Negative Control; Null hypothesis was no difference between treatments. Tests were 2-sided; Test type: Superiority or Other; p = 0.1792, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; Treatment was a fixed factor and baseline Schiff Sensitivity Score was a covariate; Adjusted mean difference = -0.12, 95% CI [-0.30 to 0.06] — Difference was calculated as adjusted mean change from baseline in 0.454% stannous fluoride toothpaste minus 0.76% sodium fluoride toothpaste. Negative difference favored stannous fluoride toothpaste

3. Secondary Outcome: Adjusted Mean Change From Baseline in Tooth Hypersensitivity to Air Stimuli at Day 14
Description: Response to a constant (duration, pressure, temperature, distance from target) jet of air applied to a hypersensitive tooth evaluated using Schiff Cold Air Sensitivity Scale. According to this analog scale hypersensitivity scores for the stimulated tooth is 0, 1, 2 or 3 (lower the score, lower the hypersensitivity). 0=No participant response to stimulus, 1=responds but will continue, 2=responds and moves or requests discontinuation, 3=Painful response to stimulus, discontinuation requested. Change was Schiff score on Day 14 minus Schiff score at baseline.
Time Frame: Baseline and Day 14
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Test: Commercially available toothpaste containing 0.454% stannous fluoride, 1 inch strip brushed on each of the 2 selected sensitive teeth for 30 seconds, followed by thorough brushing of all teeths for at least 1 minute for 14 days twice daily. The test product is a commercially available product.
Arm/Group | Test | Negative Control
Number analyzed (Participants) | 59 | 58
units on a scale | -1.24 (0.604) [-1.39 to -1.08] | -0.72 (0.622) [-0.87 to -0.56]
Statistical Analysis 1: Comparison: Test vs Negative Control; Null hypothesis was no difference between treatments. Tests were 2-sided; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; Treatment was a fixed factor and baseline Schiff Sensitivity Score was a covariate; Adjusted mean difference = -0.52, 95% CI 2-sided [-0.74 to -0.30] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Adjusted Mean Change From Baseline in Tooth Hypersensitity to Touch Stimuli (Tactile) Immediately After Treatment
Description: Measured with an electronic force sensing probe (Yeaple Probe): 10, 20, 30, 40, up to 80 grams of force applied to hypersensitive tooth until pain was elicited. Grams of force needed to elicit pain was recorded as hypersensitivity score for the tooth. The higher the score, the lower the hypersensitivity. Hypersensitivity scores on a per study participant basis was recorded as mean scores of all hypersensitive teeth. Change was calculated as mean score immediately after treatment minus mean score at baseline.
Time Frame: Baseline and immediately after treatment administration
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Test | Negative Control
Number analyzed (Participants) | 59 | 59
units on a scale | 3.73 (5.539) [2.03 to 5.43] | 3.81 (7.505) [2.11 to 5.51]
Statistical Analysis 1: Comparison: Test vs Negative Control; Null hypothesis was no difference between treatments. Tests were 2-sided; Test type: Superiority or Other; p = 0.9445, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; Treatment was a fixed factor and baseline Tactile Threshold score was a covariate; Mean adjusted difference = -0.08, 95% CI 2-sided [-2.49 to 2.32] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Adjusted Mean Change From Baseline in Tooth Hypersensitity to Touch Stimuli (Tactile) Immediately at Day 3
Description: Measured with an electronic force sensing probe (Yeaple Probe): 10, 20, 30, 40, up to 80 grams of force applied to hypersensitive tooth until pain was elicited. Grams of force needed to elicit pain was recorded as hypersensitivity score for the tooth. The higher the score, the lower the hypersensitivity. Hypersensitivity scores on a per study participant basis was recorded as mean scores of all hypersensitive teeth. Change was calculated as mean score at Day 3 minus mean score at baseline.
Time Frame: Baseline and Day 3
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Test | Negative Control
Number analyzed (Participants) | 59 | 58
units on a scale | 4.83 (7.190) [2.49 to 7.17] | 6.90 (10.630) [4.54 to 9.25]
Statistical Analysis 1: Comparison: Test vs Negative Control; Null hypothesis was no difference between treatments. Tests were 2-sided; Test type: Superiority or Other; p = 0.220, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; Treatment was a fixed factor and baseline tactile threshold score was a covariate; Adjusted mean = -2.07, 95% CI 2-sided [-5.38 to 1.25] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Adjusted Mean Change From Baseline in Tooth Hypersensitity to Touch Stimuli (Tactile) Immediately at Day 14
Description: Measured with an electronic force sensing probe (Yeaple Probe): 10, 20, 30, 40, up to 80 grams of force applied to hypersensitive tooth until pain was elicited. Grams of force needed to elicit pain was recorded as hypersensitivity score for the tooth. The higher the score, the lower the hypersensitivity. Hypersensitivity scores on a per study participant basis was recorded as mean scores of all hypersensitive teeth. Change was calculated as mean score at Day 14 minus mean score at baseline.
Time Frame: Baseline and Day 14
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Test | Negative Control
Number analyzed (Participants) | 59 | 58
units on a scale | 15.85 (12.600) [12.51 to 19.18] | 7.16 (13.249) [3.79 to 10.52]
Statistical Analysis 1: Comparison: Test vs Negative Control; Null hypothesis was no difference between treatments. Tests were 2-sided; Test type: Superiority or Other; p = 0.0004, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; Treatment was a fixed factor and baseline tactile threshold score was a covariate; Mean adjusted difference = 8.69, 95% CI 2-sided [3.96 to 13.43] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Baseline through 5 days post administration of last treatment
Groups:
- Test: Commercially available toothpaste containing 0.454% stannous fluoride, 1 inch strip brushed on each of the 2 selected sensitive teeth for 30 seconds, followed by thorough brushing of all teeth for at least 1 minute, for 14 days twice daily. The test product is a commercially available product.
Arm/Group | Test | Negative Control
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 0/59 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.